CLINICAL TRIAL: NCT06022666
Title: Application of the Palliative and Therapeutic Harmonization (PATH) Program for Shared-decision Making for Severely Frail or Cognitively Impaired Patients Scheduled for Cancer Surgery: a Randomized Control Trial.
Brief Title: PATH Program for for Severely Frail or Cognitively Impaired Patients Scheduled for Cancer Surgery.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PATHTrial
Record Dates: First submitted 2023-04-13; First posted 2023-09-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-02

CONDITIONS: Frailty; Oncology Problem; Cognitive Impairment
Keywords: frailty; cognitive impairment; cancer surgery
MeSH Terms: conditions — Frailty; Cognitive Dysfunction | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patients will undergo the usual preoperative assessment from preoperative clinic which includes standard general internal medicine and anesthesia assessment.
- PATH geriatric care (Experimental): Pre-operative assessment through the PATH clinic
  Interventions: Other: Geriatric assessment

INTERVENTIONS:
Other: Geriatric assessment — Geriatric assessment through PATH clinic which includes an evaluation of comorbidities, health trajectory and baseline frailty as well as conducting an in-depth discussion with the patient on how frailty stage impacts decision-making about surgery in order to co-develop a care plan.
  Arms: PATH geriatric care

SUMMARY:
This is a single center, non-blinded randomized control trial taking place at the Queen Elizabeth II hospital (QEII) in Nova Scotia. Patients are eligible if aged 75 and older scheduled for elective cancer surgery (proven cancer or highly suspicious cancer) and screened to have mild or greater frailty (with cognitive impairments) or moderate to greater frailty (with medical/physical conditions). Eligible participants will then be randomized to preoperative standard of care or geriatric assessment through the PATH clinic. Primary outcome will assess time spend at home at 6 months after the surgery.

DETAILED DESCRIPTION:
At Nova Scotia Health Authority (NSHA), geriatric medicine colleagues developed a preoperative palliative and therapeutic harmonization (PATH) clinic with the following objectives:

1. Assess medical conditions, health trajectory, and baseline frailty.
2. Conduct an in-depth discussion with the patient (or their substitute decision maker) to review medical conditions and how frailty stage impacts decision-making about surgery.
3. Co-develop a care plan, including ways to optimize health.

The investigators have elaborated a single center randomized cohort trial for patients aged 75 and older, screened as severely frail or cognitively impaired scheduled for curative or palliative-intent surgery for bronchopulmonary, oropharyngeal, orthopaedic, gynaecological, breast, genitourinary or gastrointestinal cancers (proven or clinically highly suspicious cancer).

Patients enrolled in the trial will be randomized to standard of care preoperative assessment versus PATH geriatric care arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a clinically highly suspicious or pathologically confirmed diagnosis of bronchopulmonary, oropharyngeal (including head and neck surgery), orthopaedic, gynaecological, breast, genitourinary or gastrointestinal cancer surgery.
2. Patients must be scheduled and consented for curative or palliative intent surgery.
3. Patients must be aged 75 or older.
4. Patients must be screened by the CFS to have:

4a. Mild or greater frailty (CFS equal or greater than 5) due to cognitive impairment.

4b. Moderate or greater frailty (CFS equal or greater than 6) due to medical/physical conditions.

5. Informed consent for participation must be received.

Exclusion Criteria:

1. Patients cannot be a resident in a long-term care facility prior to the cancer diagnosis.
2. Urgent/ emergent cases are excluded.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time spent at home 6 months following cancer surgery. | At 6 months postoperatively
  Number of days spent at home vs in a hospital or care-facility unit dichotomized as low vs high time at home. High time at home defined as 14 or fewer institution days, and low time defined as more than 14 institution days at 6 months.
Preoperative factors associated with decreased proportion of time spent at home at 6 months. | At 6 months postoperatively

SECONDARY OUTCOMES:
Number of participants requiring home care utilization | Assessed from date of hospital discharge (from index surgery) to 6 months postoperatively.
  Receipt of any homeware service (nursing, wound care, social workers, physiotherapy) from the day of postoperative discharge from the hospital.
Number of participants experiencing death or development of persistent significant new disability. | Assessed from date of index surgery to 6 months postoperatively.
  Participant passing away or developing a new disability, from the day of index surgery. Assessed using the WHODAS 2.0 disability scale.
Preoperative factors associated with increased home care utilization, death, or new onset disability. | Assessed up to 6 months postoperatively.
Rate of change to a non-operative strategy | Assessed from date of randomization until documented confirmation that patient has opted for non surgical approach, assessed up to 6 months.
  Rate of patients randomized to PATH clinic arm that end up declining surgery after consultation.
Decision regret scores. | Assessed from date of hospital discharge (from index surgery) to 6 months postoperatively.
  Decisional Regret Scale ranging from 0-100 scores measure the distress or remorse regarding the patient's decision made about undergoing surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Spence, MD, FRCSC, Principal Investigator — Queen Elizabeth II Health Sciences Center
Locations (1):
- QEII, Victoria General Hospital, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chesney TR, Coburn N, Mahar AL, Davis LE, Zuk V, Zhao H, Hsu AT, Wright F, Haas B, Hallet J; Recovery After Surgical Therapy for Older Adults Research-Cancer (RESTORE-Cancer) Group. All-Cause and Cancer-Specific Death of Older Adults Following Surgery for Cancer. JAMA Surg. 2021 Jul 1;156(7):e211425. doi: 10.1001/jamasurg.2021.1425. Epub 2021 Jul 14. PMID 33978695
- [Background] Finlayson EV, Birkmeyer JD. Operative mortality with elective surgery in older adults. Eff Clin Pract. 2001 Jul-Aug;4(4):172-7. PMID 11525104
- [Background] McIsaac DI, Taljaard M, Bryson GL, Beaule PE, Gagne S, Hamilton G, Hladkowicz E, Huang A, Joanisse JA, Lavallee LT, MacDonald D, Moloo H, Thavorn K, van Walraven C, Yang H, Forster AJ. Frailty as a Predictor of Death or New Disability After Surgery: A Prospective Cohort Study. Ann Surg. 2020 Feb;271(2):283-289. doi: 10.1097/SLA.0000000000002967. PMID 30048320
- [Background] Zhang XM, Jiao J, Xie XH, Wu XJ. The Association Between Frailty and Delirium Among Hospitalized Patients: An Updated Meta-Analysis. J Am Med Dir Assoc. 2021 Mar;22(3):527-534. doi: 10.1016/j.jamda.2021.01.065. Epub 2021 Feb 5. PMID 33549566
- [Background] Spence RT, Hirpara DH, Doshi S, Quereshy FA, Chadi SA. ASO Author Reflections: A Reductionist's Approach to Risk-Adjusted Predictions and Outcomes Assessment: Less is More. Ann Surg Oncol. 2021 May;28(5):2788-2789. doi: 10.1245/s10434-020-09284-x. Epub 2020 Nov 5. No abstract available. PMID 33151504
- [Background] Spence RT, Hirpara DH, Doshi S, Quereshy FA, Chadi SA. Will My Patient Survive an Anastomotic Leak? Predicting Failure to Rescue Using the Modified Frailty Index. Ann Surg Oncol. 2021 May;28(5):2779-2787. doi: 10.1245/s10434-020-09221-y. Epub 2020 Oct 23. PMID 33098049
- [Background] Theou O, Perez-Zepeda MU, van der Valk AM, Searle SD, Howlett SE, Rockwood K. A classification tree to assist with routine scoring of the Clinical Frailty Scale. Age Ageing. 2021 Jun 28;50(4):1406-1411. doi: 10.1093/ageing/afab006. PMID 33605412
- [Background] Hall DE, Arya S, Schmid KK, Carlson MA, Lavedan P, Bailey TL, Purviance G, Bockman T, Lynch TG, Johanning JM. Association of a Frailty Screening Initiative With Postoperative Survival at 30, 180, and 365 Days. JAMA Surg. 2017 Mar 1;152(3):233-240. doi: 10.1001/jamasurg.2016.4219. PMID 27902826
- [Background] Chesney TR, Haas B, Coburn N, Mahar AL, Davis LE, Zuk V, Zhao H, Wright F, Hsu AT, Hallet J. Association of frailty with long-term homecare utilization in older adults following cancer surgery: Retrospective population-based cohort study. Eur J Surg Oncol. 2021 Apr;47(4):888-895. doi: 10.1016/j.ejso.2020.09.009. Epub 2020 Sep 16. PMID 32980211
- [Background] Moorhouse P, Mallery LH. Palliative and therapeutic harmonization: a model for appropriate decision-making in frail older adults. J Am Geriatr Soc. 2012 Dec;60(12):2326-32. doi: 10.1111/j.1532-5415.2012.04210.x. Epub 2012 Oct 30. PMID 23110462
- [Background] Chesney TR, Haas B, Coburn NG, Mahar AL, Zuk V, Zhao H, Wright FC, Hsu AT, Hallet J; Recovery After Surgical Therapy for Older Adults Research-Cancer (RESTORE-Cancer) Group. Patient-Centered Time-at-Home Outcomes in Older Adults After Surgical Cancer Treatment. JAMA Surg. 2020 Nov 1;155(11):e203754. doi: 10.1001/jamasurg.2020.3754. Epub 2020 Nov 18. PMID 33026417